CLINICAL TRIAL: NCT04225676
Title: A Phase II, Open Label, Multi-center Trial to Determine the Efficacy and Safety of Tisagenlecleucel Re-infusion in Pediatric and Adolescent Young Adult (AYA) Patients With Acute Lymphoblastic Leukemia Experiencing Loss of B Cell Aplasia
Brief Title: Study of Efficacy and Safety of Reinfusion of Tisagenlecleucel in Pediatric and Young Adult Patients With Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019BUS03
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: CTL019; Kymriah; Tisagenlecleucel; B-Cell Acute Lymphoblastic Leukemia; Leukemia; ALL; Pediatric; Young Adult; Reinfusion
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel (Experimental): Tisagenlecleucel Cell Dispersion for Infusion given once during the study.
  The approved dose range for tisagenlecleucel is: 0.2 to 5.0×106 CAR positive viable T cells / kg for patients' ≤ 50 kg body weight or 0.1 to 2.5×108 CAR-positive viable T cells for patients > 50 kg body weight.
  Interventions: Biological: Tisagenlecleucel

INTERVENTIONS:
Biological: Tisagenlecleucel — Tisagenlecleucel Cell Dispersion for Infusion given once during the study.
  The approved dose range for tisagenlecleucel is: 0.2 to 5.0×106 CAR positive viable T cells / kg for patients' ≤ 50 kg body weight or 0.1 to 2.5×108 CAR-positive viable T cells for patients > 50 kg body weight.

SUMMARY:
This was a multi-center Phase II study investigating the efficacy and safety of reinfusion of tisagenlecleucel in pediatric and young adult patients with acute lymphoblastic leukemia (ALL) who were treated with tisagenlecleucel and experience B cell recovery.

DETAILED DESCRIPTION:
This trial was a phase II, open label, multi-center trial to determine the efficacy and safety of tisagenlecleucel re-infusion in pediatric and adolescent young adult (AYA) patients with acute lymphoblastic leukemia (ALL) experiencing loss of B cell aplasia. Loss of B-cell aplasia is defined as: peripheral blood (PB) absolute B lymphocyte count ≥ 50/µL, OR PB B lymphocyte ≥ 10% of the total lymphocytes. B-cell aplasia is defined as PB absolute B lymphocyte count <50/µL.

The study had the following phases for all patients: Screening, Treatment and Follow-up. The total duration of the study was about 12 months. After tisagenlecleucel re-infusion, efficacy was assessed at months 1, 3, 6, and End of Study at which time blood samples were obtained.

The study stopped early due to slow enrollment into the trial. The rate of enrollment made the trial no longer feasible to continue.

The patients were able to voluntarily withdraw from the study for any reason, at any time. Patients who received commercial tisagenlecleucel had to be followed for up to 15 years post-infusion. Patients could have been followed under the Center for International Blood and Marrow Transplant Research (CIBMTR) cellular therapy registry if consented for participation. For patients who do not provide consent for participation in the Center for International Blood and Marrow Transplant Research (CIBMTR) registry, adverse events were to be reported for 15 years or until the patient enrolls in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Must have an additional dose of unexpired, commercial tisagenlecleucel available and prescribed by a physician in the course of medical practice
* Age up to and including 25 years
* Patients must have CD-19+ Leukemia
* Patients who were previously treated with tisagenlecleucel and present with evidence of B-cell recovery as defined by: Peripheral blood (PB) absolute B lymphocyte count ≥ 50/µL, OR PB B lymphocyte ≥ 10% of the total lymphocytes

Exclusion Criteria:

* Prior gene therapy other than tisagenlecleucel
* Prior adoptive T cell therapy other than tisagenlecleucel
* Active CNS involvement by malignancy
* Active or latent hepatitis B or active hepatitis C, or any uncontrolled infection at screening
* HIV positive test within 8 weeks of screening

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Childrens Hospital Los Angeles Divisionof Hematology/Oncology, Los Angeles, California
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Children s Mercy Hospital, Kansas City, Missouri
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1196

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 7 participants screened.
Groups:
- Tisagenlecleucel: Tisagenlecleucel Cell Dispersion for Infusion given once during the study.
  The approved dose range for tisagenlecleucel is: 0.2 to 5.0×10^6 CAR positive viable T cells / kg for patients' ≤ 50 kg body weight or 0.1 to 2.5×10^8 CAR-positive viable T cells for patients > 50 kg body weight.
Period: Overall Study
Arm/Group | Tisagenlecleucel
Started | 5
Full Analysis, Safety and Enrolled Sets | 5
Completed | 0
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 1
Not completed — Study terminated by sponsor | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  < 10 years | 2
  >=10 to <18 years | 2
  >=18 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Establish B Cell Aplasia Within 9 Months of Reinfusion
Description: Percentage of patients who establish B-cell aplasia at any visit following re-infusion with tisagenlecleucel. B-cell aplasia is defined as peripheral blood (PB) absolute B lymphocyte count <50/μL. Planned timeframe was 12 months but actual timeframe was approximately 9 months due to early termination of the trial. Day 1 is post lymphodepleting chemotherapy and pre-reinfusion of tisagenlecleucel.
Time Frame: Post-reinfusion up to 9 months (Day 1 is excluded)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Complete Response (CR) or Complete Response With Incomplete Blood Count Recovery (CRi) by Day
Description: Overall remission rate (ORR) was defined as the percentage of participants with a best overall disease response of complete remission (CR) or CR with incomplete blood count recovery (CRi). However, the rate was not calculated due to low enrollment. Participants' best responses have been listed by day and participants may be counted more than once.
Time Frame: Post-reinfusion up to 9 months
Population: Full analysis set - Data was not adequate to perform overall remission rate analysis considering evaluable population size
Measure: Number; unit: responses
Groups:
- Complete Remission: Complete remission as determined by the investigator
- Complete Remission Without Complete Blood Count Recovery: Complete remission as determined by the investigator without complete blood count recovery
Arm/Group | Complete Remission | Complete Remission Without Complete Blood Count Recovery
Number analyzed (Participants) | 5 | 5
responses
  Day 24 | 0 | 1
  Day 28 | 1 | 0
  Day 29 | 1 | 0
  Day 32 | 1 | 0
  Day 34 | 1 | 0
  Day 67 | 1 | 0
  Day 84 | 0 | 1
  Day 91 | 0 | 1
  Day 177 | 0 | 1
  Day 182 | 1 | 0
  Day 211 | 0 | 1
  Day 274 | 0 | 1

3. Secondary Outcome: Participants With an Event
Description: An event was defined as one of the following: death from any cause after remission, relapse, treatment failure (defined as no response in the study or discontinuation from the study for death, adverse event, lack of efficacy or progressive disease or new cancer therapy).
Time Frame: Reinfusion up to 9 months
Population: Full analysis set - Data was not adequate to perform time to event analysis considering evaluable population size.
Measure: Number; unit: participant
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 5
participant | 1

4. Secondary Outcome: Overall Survival (OS)
Description: Deaths due to any reason.
Time Frame: Reinfusion up to 9 months
Population: Full analysis set - Data was not adequate to perform overall survival analysis considering evaluable population size
Measure: Number; unit: deaths
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 5
deaths | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study for a duration of 274 days. .
Arm/Group | Tisagenlecleucel
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel (N=5)
Pyrexia (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel (N=5)
Anaemia (Blood and lymphatic system disorders) | 2
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Tooth development disorder (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Catheter site erythema (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Conjunctivitis (Infections and infestations) | 1
HCoV-OC43 infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Polyomavirus viraemia (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Enterovirus test positive (Investigations) | 1
Human rhinovirus test positive (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Respirovirus test positive (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT04225676/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT04225676/SAP_001.pdf